CLINICAL TRIAL: NCT04817033
Title: Comparison of Intraoperative Complications in Patients With or Without High Risk for Obstructive Sleep Apnea During Sedation With Midazolam or Dexmedetomidine Within Transurethral Resections of Bladder and Prostate
Brief Title: Sedation Complications in Urology During Spinal Anesthesia With Dexmedetomidine or Midazolam Regarding OSA Risk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ivan Vuković, MD, Principal Investigator, University Hospital of Split
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2181-147-01/06/M.S.-20-02
Record Dates: First submitted 2021-03-18; First posted 2021-03-25 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia; Anesthesia Complication; Osa Syndrome; Transurethral Resection of Prostate; Sedation Complication; Intraoperative Complications; Snoring; Airway Obstruction
Keywords: Dexmedetomidine; Midazolam; STOP BANG questionnaire; Intraoperative complications; Spinal anesthesia; Cardiorespiratory polygraphy; sMVAP index; Sedation
MeSH Terms: conditions — Carnevale syndrome; Intraoperative Complications; Snoring; Airway Obstruction | interventions — Anesthesia, Spinal; Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: factorial randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High risk OSA Dexmedetomidine (Active Comparator): High risk OSA defined by STOP BANG questionnaire Intraoperative sedation during spinal anesthesia for transurethral resection of bladder and prostate
  Interventions: Procedure: Spinal anesthesia with intraoperative dexmedetomidine sedation; Drug: Dexmedetomidine
- High risk OSA Midazolam (Active Comparator): High risk OSA defined by STOP BANG questionnaire Intraoperative sedation during spinal anesthesia for transurethral resection of bladder and prostate
  Interventions: Procedure: Spinal anesthesia with intraoperative midazolam sedation; Drug: Midazolam
- Low&Medium OSA Dexmedetomidine (Active Comparator): Low&Medium OSA defined by STOP BANG questionnaire Intraoperative sedation during spinal anesthesia for transurethral resection of bladder and prostate
  Interventions: Procedure: Spinal anesthesia with intraoperative dexmedetomidine sedation; Drug: Dexmedetomidine
- Low&Medium OSA Midazolam (Active Comparator): Low&Medium OSA defined by STOP BANG questionnaire Intraoperative sedation during spinal anesthesia for transurethral resection of bladder and prostate
  Interventions: Procedure: Spinal anesthesia with intraoperative midazolam sedation; Drug: Midazolam

INTERVENTIONS:
Procedure: Spinal anesthesia with intraoperative dexmedetomidine sedation — Skin was disinfected and 40mg of 2% Lidocaine was given subcutaneously at lumbar vertebrae 3/4 level. 25 G spinal needle was used and after dura and arachnoidea were pierced 12.5-15 mg of 0.5% Levobupivacaine was applied.
  Arms: High risk OSA Dexmedetomidine; Low&Medium OSA Dexmedetomidine
Procedure: Spinal anesthesia with intraoperative midazolam sedation — Skin was disinfected and 40mg of 2% Lidocaine was given subcutaneously at lumbar vertebrae 3/4 level. 25 G spinal needle was used and after dura and arachnoidea were pierced 12.5-15 mg of 0.5% Levobupivacaine was applied.
  Arms: High risk OSA Midazolam; Low&Medium OSA Midazolam
Drug: Dexmedetomidine — Dexmedetomidine 0.5 ug/kg during first 10 minutes after successful spinal anesthesia. Dose maintained to keep patient in moderate sedation with closed eyes and Ramsay sedation scale 4 and 5 level
  Other Names: Dexmedetomidine sedation
  Arms: High risk OSA Dexmedetomidine; Low&Medium OSA Dexmedetomidine
Drug: Midazolam — Midazolam 0.25 mg/kg ideal body weight during first 10 minutes after successful spinal anesthesia. Dose maintained to keep patient in moderate sedation with closed eyes and Ramsay sedation scale 4 and 5 level
  Other Names: Midazolam sedation
  Arms: High risk OSA Midazolam; Low&Medium OSA Midazolam

SUMMARY:
Light to moderate sedation is recommended during surgery with spinal anesthesia . This study is exploring which sedation drug is better, midazolam or dexmedetomidine for transurethral resection of bladder and prostate in patients with or without high risk for obstructive sleep apnea (OSA). Patients were divided in two groups regarding OSA risk, and each group received midazolam or dexmedetomidine for sedation. Investigators observed intraoperative complications of airway and factors that are disturbing surgeon(movement due to participants coughing and restlessness) because one could puncture bladder or prostate and cause perforation.

DETAILED DESCRIPTION:
All participants were premedicated with diazepam 5mg 12 hours and 1 hour before surgery. Thromboprophylaxis (enoxaparin 4000-6000 IU) depending on the body weight was given at least 12 hours before surgery.

Participants were divided by STOP-BANG(Snoring history, Tired during the day, Observed stop breathing while sleep, High blood pressure, BMI more than 35 kg/m2, Age more than 50 years, Neck circumference more than 40 cm and male Gender) questionnaire into one of two groups: high OSA and low&medium OSA. Each group was then allocated by permuted block randomisation into midazolam or dexmedetomidine group. The randomisation list was obtained from R program. The group allocations were contained in closed envelope that were opened before surgery after the completed enrollment procedure.

Participants got IV cannula with switch for continuous intravenous infusion in operating theatre. Non invasive monitoring (electrodes for ECG, blood pressure cuff and pulse oximeter) was placed before induction of spinal anesthesia. Skin was disinfected and 40mg of 2% Lidocaine was given subcutaneously at lumbar vertebrae 3/4 level. 25 G spinal needle was used and after dura and arachnoidea were pierced 12.5-15 mg of 0.5% Levobupivacaine was applied. Participants were then positioned in uniform lithotomy position and 9cm pillow was inserted. After sensory block, defined as the absence of pain at T10 dermatome, was induced by needle-tip test by the anaesthesiologist, the surgery was initiated.

Time after subarachnoid block was T0 and sedation with midazolam or dexmedetomidine was started via continuous intravenous infusion. Midazolam was started with 0.25 mg/kg of ideal body mass, and dexmedetomidine with 0.5 ug/kg through 10 minutes. Every 10 minutes sedation level was observed with Ramsay sedation scale (RSS). Drug was titrated to achieve RSS of 4 or 5 (closed eyes and patient exhibited brisk or sluggish response to light glabellar tap or loud auditory stimulus). Independent blinded doctor was assessing RSS level, vital parameters and signs of airway obstruction every 10 minutes. Every 10 minutes systolic, diastolic and mean arterial pressure(MAP) were noticed along with heart rate, oxygen saturation by pulse oximetry(SpO2), RSS level and adverse intraoperative events: snoring as sign of airway obstruction, cough and restlessness as disturbing factors to surgeon. If peripheral oxygen fell below 90% supplemental oxygen was delivered by facemask with reservoir bag at flow of 10 L/min. End tidal carbon dioxide(CO2)was measured for detection of possible apnea. If oxygenation was still inadequate chin lift and jaw thrust maneuver were performed and oropharyngeal airway was inserted if needed. If heart rate fell below 50 bpm atropine 0.1 mg/kg was given and if systolic blood pressure fell below 100 mmHg(or MAP < 65 mmHg) ephedrine 5mg bolus was given. Total crystalloid infusion volume was noticed at the end of surgery. All measurements were performed every 10 minutes and 1 hour after surgery in urology intensive care. High risk OSA participants underwent cardiorespiratory polygraphy at Center for sleep medicine Split.

ELIGIBILITY:
Inclusion Criteria:

* elective transurethral resection of bladder and prostate
* American Society of Anesthesiologists (ASA) physical status classification system: I, II, III

Exclusion Criteria:

* regional anesthesia contraindications
* American Society of Anesthesiologists (ASA) physical status classification system: IV
* Atrioventricular cardiac block II and III degree
* Psychotic disorders
* Participants with tracheostomy
* Dementia
* Allergy on Dexmedetomidine or Midazolam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Airway complications | During surgery
  Snoring detection, SpO2 and patient respiration monitoring, If SpO2 fell below 90% supplemental oxygen was delivered by facemask with reservoir bag at flow of 10 L/min. If oxygenation was still inadequate chin lift and jaw thrust maneuver were performed and oropharyngeal airway was inserted.
Coughing and restlessness | During surgery
  Participants have to be relaxed and calm during surgery and sedation. Theirs coughing and restlessness result in movement that is disturbing to surgeon because they could puncture bladder/prostate with resectoscope and cause perforation. So when surgeon complains about participants movement due to theirs coughing and restlessness investigators check that on list.
Cardiorespiratory polygraphy | up to 30 weeks
  OSA classification with apnea hypopnea index(AHI) for High risk OSA participants

SECONDARY OUTCOMES:
Arterial blood pressure | During surgery
  Systolic, diastolic and mean arterial blood pressure changes, Ephedrine use if systolic blood pressure < 100 mmHg or MAP<65 mmHg
Symptomless Multi-Variable Apnea Prediction(sMVAP) index | up to 30 weeks
  OSA risk calculated by gender, age and BMI
Medications | During surgery
  Medications that participant use regularly
Heart rate | During surgery
  Atropine 0.1 mg/kg use if pulse<50
Cigarette smoking | During surgery
  Participant is active cigarette smoker or nonsmoker
ASA status | During surgery
  Participant ASA status
Crystalloid infusion | During surgery
  Volume of crystalloid infusion at the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Vukovic, Principal Investigator — University Hospital Split, Department of Anesthesiology and Intensive Care, Split, Croatia; Renata Pecotic, Study Chair — University of Split School of Medicine, Split, Croatia; Bozidar Duplancic, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care, Split, Croatia; Benjamin Benzon, Study Chair — University of Split School of Medicine, Split, Croatia; Zoran Dogas, Study Chair — University of Split School of Medicine, Split, Croatia; Ruben Kovac, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care, Split, Croatia
Locations (1):
- University Hospital Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madhusudan P, Wong J, Prasad A, Sadeghian E, Chung FF. An update on preoperative assessment and preparation of surgical patients with obstructive sleep apnea. Curr Opin Anaesthesiol. 2018 Feb;31(1):89-95. doi: 10.1097/ACO.0000000000000539. PMID 29120932
- [Background] Roesslein M, Chung F. Obstructive sleep apnoea in adults: peri-operative considerations: A narrative review. Eur J Anaesthesiol. 2018 Apr;35(4):245-255. doi: 10.1097/EJA.0000000000000765. PMID 29300271
- [Background] Corso R, Russotto V, Gregoretti C, Cattano D. Perioperative management of obstructive sleep apnea: a systematic review. Minerva Anestesiol. 2018 Jan;84(1):81-93. doi: 10.23736/S0375-9393.17.11688-3. Epub 2017 Apr 11. PMID 28402089
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Seet E, Chua M, Liaw CM. High STOP-BANG questionnaire scores predict intraoperative and early postoperative adverse events. Singapore Med J. 2015 Apr;56(4):212-6. doi: 10.11622/smedj.2015034. PMID 25917473
- [Background] Pollock JE, Neal JM, Liu SS, Burkhead D, Polissar N. Sedation during spinal anesthesia. Anesthesiology. 2000 Sep;93(3):728-34. doi: 10.1097/00000542-200009000-00022. PMID 10969306
- [Background] De Andres J, Valia JC, Gil A, Bolinches R. Predictors of patient satisfaction with regional anesthesia. Reg Anesth. 1995 Nov-Dec;20(6):498-505. PMID 8608068
- [Background] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372
- [Background] Shin HJ, Kim EY, Hwang JW, Do SH, Na HS. Comparison of upper airway patency in patients with mild obstructive sleep apnea during dexmedetomidine or propofol sedation: a prospective, randomized, controlled trial. BMC Anesthesiol. 2018 Sep 5;18(1):120. doi: 10.1186/s12871-018-0586-5. PMID 30185146
- [Background] Mingir T, Ervatan Z, Turgut N. Spinal Anaesthesia and Perioperative Anxiety. Turk J Anaesthesiol Reanim. 2014 Aug;42(4):190-5. doi: 10.5152/TJAR.2014.99705. Epub 2014 May 29. PMID 27366419